CLINICAL TRIAL: NCT05737693
Title: Posttraumatic Stress Disorder (PTSD) Treatment: Using Ketamine to Enhance Memory Reconsolidation and Extinction of Overgeneralized Fear in Individuals Diagnosed With PTSD
Brief Title: Enhancing Week-long Psychological Treatment for PTSD With Ketamine
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1509016530_a; R61MH129559 (NIH)
Record Dates: First submitted 2023-02-01; First posted 2023-02-21 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; ketamine; midazolam
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Ketamine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- 0.2mg/kg ketamine with psychotherapy (Experimental): Two infusions of low dose Ketamine combined with trauma-focused psychotherapy. Low dose ketamine infusion will take place on day 2 and day 4, of the psychotherapy intervention. A physician will oversee and administer the ketamine infusions. A nurse will accompany the subject throughout the study sessions, from the insertion of bilateral cannula for drug infusion and blood sampling, to the recovery following ketamine infusion. Whilst subjects undergo the infusion, their heart rate and blood pressure will be constantly monitored. The participant will receive a steady state of ketamine infusion of 0.2 mg/kg for 40 minutes.
  Interventions: Drug: Ketamine
- 0.5mg/kg ketamine with psychotherapy (Experimental): 2. Two infusions of Ketamine combined with trauma-focused psychotherapy. Low dose ketamine infusion will take place on day 2 and day 4, of the psychotherapy intervention. A physician will oversee and administer the ketamine infusions. A nurse will accompany the subject throughout the study sessions, from the insertion of bilateral cannula for drug infusion and blood sampling, to the recovery following ketamine infusion. Whilst subjects undergo the infusion, their heart rate and blood pressure will be constantly monitored. The participant will receive a steady state of ketamine infusion of 0.5 mg/kg for 40 minutes.
  Interventions: Drug: Ketamine
- Midazolam with psychotherapy (Active Comparator): Midazolam combined with trauma-focused psychotherapy. Midazolam infusion procedure will take place on day 2 and day 4, of the psychotherapy intervention. A physician will oversee administer the Midazolam infusions. A nurse will accompany the subject throughout the study sessions, from the insertion of bilateral cannula for drug infusion and blood sampling, to the recovery following midazolam infusion. Whilst subjects undergo the infusion, their heart rate and blood pressure will be constantly monitored. The participant will receive a steady midazolam infusion at a rate 0.045 mg/kg for 40 minutes.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Ketamine — Week-long exposure therapy with ketamine infusion on day 2 and 4 of the psychotherapy
  Other Names: Ketalar
  Arms: 0.2mg/kg ketamine with psychotherapy; 0.5mg/kg ketamine with psychotherapy
Drug: Midazolam — Week-long exposure therapy with midazolam infusion on day 2 and 4 of the psychotherapy
  Other Names: Versed
  Arms: Midazolam with psychotherapy

SUMMARY:
The purpose of this study is to test if the combination of ketamine, vs midazolam, with an intensive trauma-focused psychotherapy will be more effective in relieving post-traumatic stress disorder (PTSD). This week-long treatment has the potential to produce a significant therapeutic effect that otherwise would take months to occur. The study will also focus on learning about the neurophysiological changes produced by the proposed clinical trial.

DETAILED DESCRIPTION:
Based on the current research findings on the therapeutic effectiveness of trauma focus psychotherapy and of ketamine combining the two treatments may yield a promising new rapid week-long treatment for PTSD. As PTSD symptoms' structure is comprised of several unique clusters which include re-experiencing, avoidance, depression and hypervigilance the investigators hypothesize that by combining Ketamine with trauma-focused psychotherapy the proposed intervention can address these PTSD symptoms clusters more effectively than existing treatments. This proposed clinical trial has the potential to produce a significant therapeutic effect that otherwise would take months to occur by tapping on the enhanced neuroplasticity and the antidepressant effect of ketamine (which lasts between 24hrs to 7 days), to promote rapid changes in learning and memory when applying psychotherapy within a unique "window of opportunity" of neurophysiological changes produced by the investigative drug.

During the first visit participants will undergo a clinical interview to establish a PTSD diagnosis and other eligibility criteria. If found eligible participants will be invited to take part in this 7-day rapid treatment trial for PTSD.

On the first therapy visits, participants will be educated about the psychological treatment that will be provided and the potential benefit of ketamine or midazolam that may enhance the psychotherapy outcomes.

On the second day of the study, participants will receive an infusion of ketamine or midazolam and will undergo a magnetic resonance imaging (MRI) to assess their brain reactivity to PTSD before the treatment.

On days 3-6 participants will attend a 60-90 minutes psychotherapy session to address their PTSD symptoms.

A second ketamine or midazolam infusion will take place on day 4 of the study to enhance the drug therapeutic effect for the study duration.

Day 7 will include another MRI scan to assess treatment effect on PTSD.

Participants will need to attend one follow up MRI scan and clinical evaluation at 30 days and then a clinical evaluation at 90 days post-treatment to assess the long-term effectiveness of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 21-70 years. This age range was chosen to fit with prior samples in which no adverse effects of ketamine have been observed. Adults in the 18-20 ranges have been eliminated because previous experience indicates that they often lack the maturity to participate effectively in similar protocols. Females will be included if they are not pregnant and agreed to utilize a medically accepted birth control method (to include oral, injectable, or implant birth control, condom, diaphragm with spermicide, intrauterine device, tubal ligation, abstinence, or partner with vasectomy) or if post-menopausal for at least 1 year, or surgically sterile.
* Must not have a medical/neurological problem or use medication that would render ketamine unsafe by history or medical evaluation.
* Diagnosis of chronic PTSD with a score of 25 or higher (i.e. severe PTSD) on the Clinician-Administered PTSD Scale (CAPS-5) at screening. PTSD symptoms must have persisted for >1 year post-trauma exposure to meet the DSM-5 definition of chronic.
* Subjects on FDA-approved antidepressant, trazodone, atypical neuroleptic, prazosin, or clonidine may enter the study if they have been on a stable treatment, as determined by the study clinician, for at least 4 weeks prior to randomization. Following randomization, small changes to doses may be allowable at the PI's discretion.
* Able to provide written informed consent.
* Able to read and write English.

Exclusion Criteria:

* Patients with a diagnostic history of borderline personality disorder, obsessive compulsive disorder, schizophrenia or schizoaffective disorder or currently exhibiting psychotic features as determined by the Structured Clinical Interview for DSM (SCID); dementia or suspicion thereof, are excluded. Patients with history of bipolar disorder will be included only if they have not experienced a manic or hypomanic episode in the 30 days prior to enrollment. Other DSM Axis I disorders are permitted as long as they are not considered primary disorders.
* Patients with a history of antidepressant-induced hypomania or mania as determined by open-ended psychiatric interview.
* Current, ongoing serious suicidal risk as assessed by evaluating investigator based on the Columbia-Suicide Severity Rating Scale (C-SSRS).
* Moderate severity or greater Substance Use Disorder (excepting Alcohol and Marijuana Use Disorder) during the 3 months prior to randomization, as determined by the SCID.Alcohol or Marijuana Use Disorder may be allowed based on the judgment of study physician/APRN/clinician that patients can remain sober for all study visits.
* Subjects on a prohibited medication (see Table 1). Patients will not be taken off medication for the purpose of this study.
* History of traumatic brain injury (TBI) with loss of consciousness for more than 24 hours or posttraumatic amnesia for more than 7 days may be considered if the trauma occurred more than 1 year ago, and no more than minimal symptoms have persisted over the past year.
* Positive pregnancy test at screening or prior to any study drug infusion.
* Breathalyzer showing an alcohol level > 0% at screening, or at the discretion of the investigator, prior to any study drug infusion.
* Resting blood pressure lower than 90/60 or higher than 150/90, or resting heart rate lower than 45/min or higher than 100/min.
* Any significant history of serious medical or neurological illness.
* Any signs of major medical or neurological illness on examination or as a result of ECG screening or laboratory studies.
* Abnormality on physical examination. A subject with a clinical abnormality may be included only if the study physician considers the abnormality will not introduce additional risk factors and will not interfere with the study procedure.
* A positive pre-study (screening) urine drug screen or, at the study physician's discretion on any drug screens given before the scans.
* Pregnant or lactating women or a positive urine pregnancy test for women of child-bearing potential at screening or prior to any imaging day.
* Any history indicating learning disability or mental retardation.
* Known sensitivity to ketamine.
* Body circumference of 52 inches or greater.
* Body weight of 350 pounds or greater.
* History of claustrophobia.
* Presence of cardiac pacemaker or other electronic device or ferromagnetic metal foreign bodies in vulnerable positions as assessed by a standard pre-MRI screening questionnaire.
* Donation of blood in excess of 500 mL within 56 days prior to dosing.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Active engagement in trauma-focused CBT (TF cognitive-behavioral therapy) or any evidence-based PTSD psychotherapy (CPT, PE, EMDR) initiated within the past 3 months (continuation of established maintenance supportive therapy will be permitted
* Enrollment in another research study testing an experimental/clinical/behavioral intervention intended to affect symptoms initiated within the last 2 months, or intended enrollment within the next 3 months

Table 1. Concomitant Treatments that are prohibited

MAOIs: 4-weeks off medication prior to randomization is required.

Memantine: 4-weeks of medication prior to randomization is required.

Long Acting Benzodiazepines -Chlordiazepoxide, Diazepam, Flurazepam: 2-weeks off medication prior to randomization is required.

Notes: As above, individuals who have used any of the prohibited medications within the "weeks off" time period will not be eligible for the study. Use of sedatives, hypnotics, benzodiazepines, sedating antihistamines or other psychotropic medications are not permitted within 8 hours of treatment sessions; except - at the discretion of the investigator - for medications that will result in discontinuation/withdrawal symptoms or that may alter the risk benefit ratio.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2030-08-01 (Estimated); Study Completion 2031-08-01 (Estimated)

PRIMARY OUTCOMES:
Amygdala activation to trauma memory (Phase 1; R61) | Changes from baseline to 30-day post-treatment in amygdala activation to the trauma memory
  Phase 1 (R61) investigators will analyze the first 60 participants (20 per arm). Using MRI scan data, the investigators will compare changes in the amygdala bold activation from baseline to 30-day post treatment in response to the trauma scripts between the the 3 study arm. Greater activation of the amygdala is an indicator of a greater distress.
  Investigators will also measure the effect size resulting from the mean changes in amygdala activation from pre to post treatment between each of the experimental groups and the active comparator to determine the dose that will be carried to phase 2.
To determine if ketamine + exposure therapy results in clinical improvement in PTSD symptoms which are significantly greater than midazolam + exposure therapy (Phase 2; combined R61/R33 data) | Baseline, 7 days, 30 days and 90 days
  Change in PTSD symptoms from baseline up to 90-day post treatment. PTSD Symptoms severity will be evaluated overtime using PTSD Check List (PCL-5).
  Evidence for the PCL suggests that 10 points difference in the measure is a reliable indicator for a clinically meaningful change. The PCL scores ranges from 0 (no symptoms) to a maximum score of 80 (PCL Score > 33 indicates probable PTSD diagnosis).
To determine if ketamine + exposure therapy results in more profound changes in task-based connectivity in region of interest than midazolam + exposure therapy (Phase 2; combined R61/R33 data) | Baseline, 7 days and 30 days (no MRI scan at 90 days post-treatment)
  Using MRI brain activation data, the investigators will compare changes in the connectivity between participants' different brain regions (brain network connectivity) from baseline to end of treatment and 30-day post treatment. Investigators will examine the neural connectivity between the amygdala, hippocampus, prefrontal cortex, striatum and insula and other major brain areas associated with PTSD.

SECONDARY OUTCOMES:
Change from baseline to 90 days post treatment in Beck Depression Inventory (BDI-II) | Baseline, 7 days, 30 days and 90 days
  The self-report BDI-II will be used to assess severity of depressive symptoms. A higher score is associated with higher severity of depression. The score is interpreted as follows: 0-13 indicates minimal depression, 14-19 indicates mild depression, 20-28 indicates moderate depression and 29-63 indicates severe depression
Measure the changes in psychophysiological distress to trauma reminders as a result of the proposed intervention | Baseline, 7 days and 30 days
  Using wrist mobile galvanic skin responses (GSR) device the investigators will measure changes in GSR from pre to post treatment during exposure to avoidance cue. Investigators will compare the magnitude of these changes between the study arms. Higher GSR indicate a greater level of distress.

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Harpaz-Rotem, PhD ABPP, Principal Investigator — Yale University
Locations (2):
- Yale University School of Medicine, New Haven, Connecticut, United States
- Tel Aviv University, Tel Aviv, Israel

DOCUMENTS (1):
  • Informed Consent Form (2023-09-05): https://cdn.clinicaltrials.gov/large-docs/93/NCT05737693/ICF_000.pdf